CLINICAL TRIAL: NCT02245620
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Impact of a Single Intravenous Dose of MTP-131 (Bendavia™) on Skeletal Muscle Function in the Elderly
Brief Title: A Phase 2 Study to Evaluate the Impact of MTP-131 (Bendavia™) on Skeletal Muscle Function in Elderly
Acronym: MOTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPITM-201
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Skeletal Muscle Mitochondrial Dysfunction in the Elderly
Keywords: Skeletal muscle dysfunction, MTP-131, Bendavia™; elamipretide
MeSH Terms: interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elamipretide (Experimental): Elamipretide given as an intravenous infusion of 0.25 mg/kg/hr at a rate of 60 mL/hr for 2 hours.
  Interventions: Drug: Elamipretide
- Placebo (Placebo Comparator): Placebo (lyophilized excipients without elamipretide) given as an intravenous infusion at a rate of 60 mL/hr for 2 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elamipretide — Elamipretide 0.25 mg/kg/hour administered as an intravenous infusion at the rate of 60 mL/hour for 2 hours
  Other Names: MTP-131; Bendavia™
  Arms: Elamipretide
Drug: Placebo — Placebo administered as intravenous infusion at a rate of 60 mL/hour for 2 hours
  Other Names: elamipretide
  Arms: Placebo

SUMMARY:
This was a Phase 2, randomized, double-blind, placebo-controlled study, enrolling 41 elderly subjects with previous evidence of mitochondrial dysfunction to evaluate whether the administration of MTP-131 (elamipretide) will change either hand skeletal muscle energetics or muscle performance in age-related skeletal muscle mitochondrial dysfunction.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, double-blind, placebo-controlled study, enrolling 41 elderly subjects with previous evidence of mitochondrial dysfunction to evaluate whether the administration of MTP-131 (elamipretide) will change either hand skeletal muscle energetics or muscle performance in age-related skeletal muscle mitochondrial dysfunction.

Subjects were randomized 1:1 to receive either elamipretide at 0.25 mg/kg/hr intravenously at a rate of 60 mL/hr for 2 hours, or placebo (lyophilized excipients without elamipretide) intravenously at a rate of 60 mL/hr for 2 hours. Each treatment group went through three distinct periods: Screening (up to 28 days), Treatment (1day), and Observation (7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Are male and female adults aged ≥60 and ≤85 years
2. Female subjects must be post-menopausal
3. Have in vivo phosphorus-31 (31P) Magnetic Resonance Spectroscopy (MRS) and (Optical Spectra Scan (OPS) determined maximum adenosine triphosphate synthetic rate (ATPmax) < 0.70 milliMol/second (mM/sec)
4. Have in vivo 31P MRS and OPS determined P/O (Phosphate/Oxygen ratio) < 1.9
5. Are ambulatory and able to perform activities of daily living without assistance
6. Had sufficient venous access for study drug administration and clinical testing.
7. Could speak and read English fluently.
8. Provided informed consent.

Exclusion Criteria:

1. Had significant disease(s) or condition(s) which, in the opinion of the Investigator, may have put the subject at risk because of their participation in the study or may have influenced either the results of the study or the subject's ability to participate in the study.
2. Had a history of rhabdomyolysis.
3. Had been hospitalized within 3 months prior to Screening for major atherosclerotic events (e.g., myocardial infarction, target-vessel revascularization, coronary bypass surgery or stroke) or other major medical condition (as deemed by the Primary Investigator).
4. Had any metal implants that could not be removed from the body that in the opinion of the Investigator were a contra-indication for undergoing the MRS procedure or any other protocol-related procedure.
5. Had an implanted cardiac pacemaker or other implanted cardiac device.
6. Had a serum sodium level <136 milliequivalents per litre (mEq/L) at Screening or Pre-infusion.
7. Had a hemoglobin level <12 g/dL at Screening or Pre-infusion.
8. Had chronic, uncontrolled hypertension as judged by the Investigator (e.g., Baseline systolic blood pressure [SBP] >140 mm Hg, diastolic blood pressure [DBP] > 90 mm Hg) or a SBP >150 mm Hg or DBP >95 mm Hg at the time of Screening or Baseline (if the initial blood pressure [BP] reading was above these values, the reading may have been repeated one time within 20 minutes of the initial reading).
9. Had a body mass index (BMI) of <16 or >35 kg/m2.
10. Had a creatinine clearance <45 mL/min as calculated by the Cockcroft Gault equation.
11. Had a 12-lead electrocardiogram (ECG) demonstrating severe bradycardia (heart rate < 40 bpm) or average corrected QC interval (QTc) >450 ms for males and > 470 ms for females, and in the opinion of the Investigator was clinically significant. (If on the initial ECG, QTc exceeded 450 ms for males or 470 ms for females, the ECG was to be repeated 2 more times and the average of the 3 QTc values was to be used to determine the subject's eligibility).
12. Had a neurologic disorder that in the opinion of the Investigator was a contra-indication for enrollment into the study.
13. Had any symptoms consistent with or a current diagnosis of peripheral neuropathy, such as numbness, tingling, pain, or altered sensation of hands or feet.
14. Had an active, systemic autoimmune disease other than autoimmune thyroid disease (e.g., diabetes, lupus, rheumatoid arthritis) that currently required treatment or was likely to require treatment during the study.
15. Subject's right hand had a history of mobility impairment, fractures, arthritis, hand surgery, muscle disease or other injury that may interfere with any study procedure.
16. Had any symptoms consistent with or a current diagnosis of claustrophobia.
17. Had a history of cancer, unless subject had documentation of completed curative treatment.
18. Had a history of or risk factors (e.g., significant family history, concomitant medical condition) for deep vein thrombosis or pulmonary embolism.
19. Had a history of serious mental illness as judged by the Investigator.
20. Had a body temperature > 37.5°C at the time of planned dosing.
21. Subjects who in the opinion of the Investigator abused alcohol or drugs.
22. Had donated or received blood or blood products within the past 30 days.
23. Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family was defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
24. Sponsor employees and/or their immediate families. Immediate family was defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
25. Were currently enrolled in a clinical study involving an investigational product or non-approved use of a drug or device or concurrently enrolled in any other type of medical research judged to be scientifically or medically incompatible with this study.
26. Had participated, within the last 30 days, in a clinical study involving an investigational product. If the previous investigational product had a long half-life, 3 months or 5 half-lives (whichever was longer) should have passed.
27. Had previously been randomized into any study investigating elamipretide or been exposed to elamipretide for any reason.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Carr, Study Director — Stealth BioTherapeutics
Locations (1):
- The University of Washington Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects discontinued prematurely as per Investigator's discretion. These 2 subjects (Subject 001019 [Elamipretide group] and Subject 001063 [Placebo group]) were discontinued after randomization but prior to receiving study treatment; both were not treated due to their pre-infusion sodium levels meeting Exclusion Criteria 6.
Groups:
- Elamipretide: Elamipretide administered as an intravenous infusion of 0.25 mg/kg/hr at a rate of 60 mL/hr for 2 hours.
Period: Overall Study
Arm/Group | Elamipretide | Placebo
Started | 20 | 21
Completed | 19 | 20
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- MTP-131 (Bendavia™): MTP-131 (Bendavia™) administered as an intravenous infusion of 0.25 mg/kg/hr at a rate of 60 mL/hr for 2 hours.
- Total: Total of all reporting groups
Arm/Group | MTP-131 (Bendavia™) | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (3.35) | 69.0 (3.96) | 68.5 (3.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 8 | 13 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39
Body Mass index [Mean (Standard Deviation); unit: kg/m²] | 26.5 (4.27) | 26.1 (2.82) | 26.3 (3.56)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ATPmax (Maximal ATP Synthetic Rate)
Description: Maximal ATP synthetic rate (phosphorylation capacity per unit muscle volume) as determined by a muscle fatigue test.
Time Frame: From Baseline, Day 1 Hour 2 (2 hours after the start of infusion, or end of infusion) and Day 7
Population: All participants for whom Maximal ATP synthetic rate was measured at baseline and Day 1 Hour 2, and Day 7
Measure: Mean (Standard Deviation); unit: mM/sec
Arm/Group | MTP-131 (Bendavia™) | Placebo
Number analyzed (Participants) | 19 | 20
mM/sec
  Day 1 Hour 2: number analyzed (Participants) | 18 | 19
  Day 1 Hour 2 | 0.17 (0.196) | 0.12 (0.244)
  Day 7 | 0.09 (0.142) | 0.06 (0.172)

2. Secondary Outcome: Mean Change From Baseline in Phosphate/Oxygen (P/O) Ratio
Description: As a measure of mitochondrial hand skeletal muscle energetics, mitochondrial coupling, or Phosphate/Oxygen ratio (P/O) was assessed at Baseline, Day 1 Hour 2, and Day 7.
Time Frame: From Baseline, Day 1 Hour 2 (2 hours after the start of infusion, or end of infusion) and Day 7
Population: All participants for whom Phosphate/Oxygen (P/O) ratio was measured at baseline and Day 1 Hour 2, and Day 7
Measure: Mean (Standard Deviation); unit: ratio of phosphate to oxygen
Arm/Group | MTP-131 (Bendavia™) | Placebo
Number analyzed (Participants) | 19 | 20
ratio of phosphate to oxygen
  Day 1 Hour 2: number analyzed (Participants) | 18 | 20
  Day 1 Hour 2 | 0.25 (0.679) | 0.26 (0.693)
  Day 7 | 0.32 (0.473) | 0.51 (0.788)

3. Secondary Outcome: Mean Change From Baseline in Nicotine Adenine Dinucleotide (NAD)
Time Frame: From Baseline, Day 1 Hour 2 (2 hours after the start of infusion, or end of infusion) and Day 7
Population: All participants for whom Nicotine Adenine Dinucleotide (NAD) was measured.
Measure: Mean (Standard Deviation); unit: millimolar
Arm/Group | MTP-131 (Bendavia™) | Placebo
Number analyzed (Participants) | 19 | 20
millimolar
  Day 1 Hour 2: number analyzed (Participants) | 18 | 20
  Day 1 Hour 2 | 0.04 (0.169) | 0.01 (0.213)
  Day 7 | 0.11 (0.215) | 0.09 (0.263)

4. Secondary Outcome: Mean Change From Baseline in Muscle Force-Time-Integral (FTI)
Description: Muscle Force-Time-Integral was measured as mean change from baseline at Day 1 Hour 2, Day 3, and Day 7.
Time Frame: From Baseline to Day 1 Hour 2, Day 3, and Day 7
Population: All participants for whom Muscle Force-Time-Integral (FTI) was measured.
Measure: Mean (Standard Deviation); unit: Newton/second
Arm/Group | MTP-131 (Bendavia™) | Placebo
Number analyzed (Participants) | 19 | 20
Newton/second
  Day 1 Hour 2 | 0.43 (0.882) | 0.10 (0.728)
  Day 3: number analyzed (Participants) | 18 | 20
  Day 3 | 0.46 (1.036) | 0.24 (0.948)
  Day 7 | 0.83 (1.485) | 0.44 (1.114)

ADVERSE EVENTS:
Time Frame: 36 days
Arm/Group | Elamipretide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 3/19 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elamipretide (N=19) | Placebo (N=20)
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less